CLINICAL TRIAL: NCT05680571
Title: Validation of Bulbicam for Use on Patient Suffering From Parkinson and Ataxia
Brief Title: Validation of Bulbicam for Parkinson- and Ataxia-patients
Status: Completed | Type: Observational
Sponsor: Meddoc (Other)
Responsible Party: Principal Investigator, Prof Stig Larsen, Professor, Meddoc
Other Study IDs: V3-NEU/PD; Ataxia-I/2022
Record Dates: First submitted 2022-07-01; First posted 2023-01-11 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Parkinson Disease; Ataxia
MeSH Terms: conditions — Parkinson Disease; Ataxia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Parkinson: Patients suffering from PD of both genders above 18 years of age and Gender- and age-matched HC without any eye- or neurological disorder.
  Interventions: Device: BulbiCam
- Ataxia: Patients suffering from AT of both genders above 18 years of ageand Gender- and age-matched HC without any eye- or neurological disorder.
  Interventions: Device: BulbiCam

INTERVENTIONS:
Device: BulbiCam — BulbiCam is an non-invasive, multi-test device which combined eye tracking; pupil metric; video graphic dual device including the f10 tests under development and ready for validation

SUMMARY:
Aim is to investigate repeatability and stability of four Neurological-related Bulbicam tests in patients suffering Parkinson (PD),Ataxia (AT) and matched healthy control (HC).

Study population The study consists of the patients suffering from PD or AT and HV of both genders above 18 years of age without any eye- or neurological disorder.

Bulbicam will be used in the study and five tests will be performed

The study will be performed as a controlled, open and non-randomized, stratified observational single center. The stratification factors will be pathology (PD&AT) and internal classifications. ed.

The main variables will be the variables recorded at the four Bulbicam tests and the standard neuro-ophthalmological variables included for PD and AT

Participants, who fulfil the inclusion criteria; do not meet any of the exclusion criteria and willing to give informed consent to participate will receive an appointment for starting the study. During the first day of the study, the included patients will undergo a neuro-ophthalmological examination by a neurologist. Additionally, Bulbicam examination will be performed twice with a rest period of one hour between each registration.

The healthy controls will only undergo a standard examination and twice BulbiCam examination. The controls will only participate one day. The patients will participate two more days with two Bulbicam examinations per day.

Sample size:

Sixteen PD-patients ,16 AT-patients and 32 HCs will be included in the study.

DETAILED DESCRIPTION:
Aim

* To investigate repeatability and stability of four Neurological-related Bulbicam tests in patients suffering from PD, AT and HC.
* To contribute to establishment of normal range for PD and AT patients with different degree in the disease development related to the Bulbicam tests.
* To contribute to establishment of normal range of these Bulbicam tests for a normal population without neurological or ophthalmological disease.

Study population The study consists of the following three study populations: 1) Patients suffering from PD of both genders above 18 years of age; 2) Patients suffering from AT of both genders above 18 years of age; 3) Gender- and age-matched HC without any eye- or neurological disorder.

Trial equipment Bulbicam will be used in the study and the following five tests will be performed at each investigation: "Fixation", "Saccade" "Nystagmus", "Smooth pursuit" and "Pupil".

Design:

The study will be performed as a controlled, open and non-randomized, stratified observational single center. The stratification factors will be pathology (PD&AT) and internal classifications. Within each of the two basic strata, healthy matched controls related to gender and age (1:1) will be included. No internal classification will be used for PD, but AT will be stratified in:

1. Patients with Nystagmus
2. Patients without Nystagmus For each included patient, a gender- and age-matched HV will be included.

The main variables will be the variables recorded at the four Bulbicam tests. The standard neuro-ophthalmological variables included for PD and AT are Nystagmus, Smooth pursuit and Saccade Accurate.

Study procedure:

Participants, who fulfil the inclusion criteria; do not meet any of the exclusion criteria and willing to give informed consent to participate will receive an appointment for starting the study. During the first day of the study, the included patients will undergo a neuro-ophthalmological examination by a neurologist. Additionally, Bulbicam examination will be performed twice with a rest period of one hour between each registration.

The healthy controls will only undergo a standard examination and twice BulbiCam examination. The controls will only participate one day. The patients will participate two more days with two Bulbicam examinations per day.

All demographic data, social factors and history of disease will be recorded at screening. The general quality of life (QoL) questionnaires EQ-5D-5L developed by EuroQol will be recorded initially as individual baseline values.

The Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be used for measuring and classifying the tolerability and toxicity at the end of each day of investigation.

Sample size:

Sixteen PD-patients and 16 AT-patients, equally divided between the internal pairs of strata, will be recruited from the participating hospital. For each included patient, one gender- and age-matched HC will be recruited. In total of 32 HC, 16 PD and 16 AT patients will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with either PD or AT of both gender; at least the age of 18 years; without any other eye disease; suffering from other know serious disease but have a health situation in accordance with expectations related to the age.
* gender- and age-matched controls to patients ; passed the age of 18 years without any eye diseases; not suffering from other know serious disease and have a health situation in accordance with expectations related to the age.

Exclusion Criteria:

* Other visual disturbances and blindness
* Posterior Chamber Intraocular Lens (PCIOL)
* Physical or psychiatric disease, which may disturb the measuring procedure
* Paresis or paralysis of any oculomotor muscle
* Patients whose visual acuity is less than 0.1 in any eye, as these will not be able to focus on the test stimuli.
* Patients whose visible part of the eye is abnormal, such as subconjunctival haemorrhages or deformed pupils
* Patients whose pupils are not able to respond normally to dilation or contraction due to damaged nerves, mechanical damage of the pupil etc.
* With known alcoholic and drug dependency
* Not able to understand information.
* Not willing to give written consent to participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of PD and AT-patients of both gender; past the age of 18 years; without any other eye disease and suffering from other know serious disease, but have a health situation in accordance with expectations related to the age.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2022-12-19 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Nystagmus | 1 hour
  Frequency in Hz
Nystagmus | 2 hours
  Frequency in Hz
Nystagmus | 24 hours
  Frequency in Hz
Nystagmus | 25 hours
  Frequency in Hz
Nystagmus | 36 hours
  Frequency in Hz
Nystagmus | 37 hours
  Frequency in Hz
Fixation | 1 hour
  Stability in mm
Fixation | 2 hours
  Stability in mm
Fixation | 24 hours
  Stability in mm
Fixation | 25 hours
  Stability in mm
Fixation | 36 hours
  Stability in mm
Fixation | 37 hours
  Stability in mm
Smooth pursuit 1 | 1 hour
  Gain velocity in degree
Smooth pursuit 1 | 2 hours
  Gain velocity in degree
Smooth pursuit 1 | 24 hours
  Gain velocity in degree
Smooth pursuit 1 | 25 hours
  Gain velocity in degree
Smooth pursuit 1 | 36 hours
  Gain velocity in degree
Smooth pursuit 1 | 37 hours
  Gain velocity in degree
Saccade | 1 hour
  Latency in ms
Saccade | 2 hours
  Latency in ms
Saccade | 24 hours
  Latency in ms
Saccade | 25 hours
  Latency in ms
Saccade | 36 hours
  Latency in ms
Saccade | 37 hours
  Latency in ms
Pupil | 1 hour
  Diameter in mm
Pupil | 2 hours
  Diameter in mm
Pupil | 24 hours
  Diameter in mm
Pupil | 25 hours
  Diameter in mm
Pupil | 36 hours
  Diameter in mm
Pupil | 37 hours
  Diameter in mm

CONTACTS AND LOCATIONS:
Overall Officials: Emilia Kerty, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
No plan